CLINICAL TRIAL: NCT05908383
Title: Phase I Clinical Study on the Safety, Tolerability and Pharmacokinetic Characteristics of a Single Dose of GMDTC Administered to Healthy Subjects for Injection
Brief Title: Safety Study of GMDTC Injection in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jianersheng (Zhuhai) Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: JianerShengPharmaTC
Record Dates: First submitted 2023-05-30; First posted 2023-06-18 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Cadmium Exposure
Keywords: cadmium; Cadmium Poisoning; Therapeutics; Drugs, Investigational
MeSH Terms: conditions — Cadmium Poisoning | interventions — Injections; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This clinical study is a double-blind study, in which participants such as clinical researchers, project managers, and project monitors are unaware of the random coding and drug administration groups of the subjects. Non-blind monitoring during the clinical study will be conducted by non-blind monitors. In addition, drug preparation will be carried out by non-blind researchers independent of this study. Analysis and testing personnel will also adopt blind analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GMDTC for injection (Experimental): The subjects assigned to the treatment group will receive once medication at 8:00 am on the second day after admission.
  Interventions: Drug: GMDTC for injection
- Normal saline group (Placebo Comparator): The subjects assigned to the placebo group will receive once medication at 8:00 am on the second day after admission.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: GMDTC for injection — GMDTC for injection with a specification of 0.5g/vial, 250mg,500mg,850mg,1200mg,1600mg,2000mg, and administered by intravenous infusion. Using 0.9% physiological saline (0.5g will be prepared with 250mL injection solution to achieve a concentration of 2mg/mL). Using an infusion pump at a rate of 4mL/min according to the dosage, and any infusion reactions will be recorded. The injection solution for both the experimental and placebo groups should be prepared by a non-blind investigator independent of the trial.
  Other Names: GMDTC Group
  Arms: GMDTC for injection
Other: Normal saline — 0.9% physiological saline for injection with a specification of 250ml/bag, and administered by intravenous infusion. Using an infusion pump at a rate of 4mL/min according to the dosage, and any infusion reactions will be recorded. The injection solution for both the experimental and placebo groups should be prepared by a non-blind investigator independent of the trial.
  Other Names: Normal saline Group
  Arms: Normal saline group

SUMMARY:
This trial is a randomized, double-blind, single-center, single-dose escalating Phase I clinical trial designed to evaluate the safety, tolerability, and pharmacokinetic characteristics of injectable GMDTC in healthy subjects

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of a single dose of injectable GMDTC in healthy subjects and to determine the maximum tolerated dose (MTD). The secondary objective is to evaluate the pharmacokinetic characteristics of injectable GMDTC after a single dose in healthy subjects and its impact on cadmium levels in the body.The modified Fibonacci method (also known as the Fibonacci dose escalation method) was used for dose escalation, with six predetermined dose groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, both male and female are eligible;
* Male subjects must weigh at least 50.0 kg and female subjects must weigh at least 45.0 kg, with a body mass index (BMI) between 19 and 26 kg/m2, including the critical value;
* Subjects must voluntarily sign a written informed consent form.

Exclusion Criteria:

* past or current clinical significant diseases that affect the circulatory, endocrine, nervous, digestive, respiratory, renal, hematological, immunological, psychiatric, and metabolic systems or any other disease or symptom that may interfere with the study results;
* eGFR<90 mL/min/l.73 m2 during screening (eGFR calculated using the Cockcroft-Gault formula: eGFR (mL/min/1.73 m2) =*(140-age)weight (kg)/[0.818Cr (umol/L)]*0.85 (female));
* urine creatinine (Cr) > 5 umol/mol for two consecutive days during screening (with a creatinine concentration of≥0.3 g/L and ≤3 ug/L);
* a history of allergy to drugs, food, or other substances, especially to the components of the study drug;
* undergone or planned surgery that affects drug metabolism and safety assessment within 4 weeks before screening;
* use of any medication or health supplements (including Chinese herbal medicine) within 14 days before screening;
* participated in any clinical trial and used any investigational drug within three months before screening;
* blood donation or significant blood loss (≥200 mL, excludingmenstrual bleeding in women) within 3 months before screening, blood transfusion, or use of blood products;
* inability to tolerate venipuncture and/or history of fainting or needle phobia;
* pregnant or lactating women, and subjects who cannot adopt effective non-drug contraceptive measures during the study period;
* unable to adopt contraceptive measures within 6 months after the end of the study;
* have special dietary requirements and cannot adhere to a uniform diet;
* daily consumption of excessive tea, coffee, and/or caffeine-containing beverages (more than 8 cups, 1 cup - 250 mL);
* unable to stop using any tobacco products during the study period;
* alcoholics or frequent drinkers within 6 months before screening, i.e., drinking more than 14 units of alcohol per week (1 unit - 360.5 mL of beer or 45 mL of 40% alcohol or 150 mL of wine) or unable to stop using any alcohol-containing products during the study period;
* drug abusers or those who used soft drugs (such as marijuana) within 3 months before screening or used hard drugs (such as cocaine, benzoyl peroxide, etc.) within 1 year before screening;
* clinically significant abnormalities in vital signs, physical examination, electrocardiogram, electroencephalogram, cardiac ultrasound, abdominal ultrasound, chest CT, ophthalmic examination, or laboratory tests (as judged by the clinical research physician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Adverse events | Up to 30 days
  Adverse events will be evaluated according to the NCI Common Terminology Criteria for Adverse Events (CTCAE, V5.0), which includes spontaneously reported adverse events as well as clinically significant changes in vital signs, physical examination, laboratory tests, electrocardiogram, and other examinations conducted during the trial.
DLT | up to 1 weeks
  DLT is defined as the occurrence of any of the following adverse events defined by NCI CTCAE V5.0 after drug administration: 1) grade 3 (severe) toxicity related to the investigational drug, such as events resulting in hospitalization or leading to serious or permanent disability or defect; 2) grade 4 (life-threatening) toxicity or any toxicity deemed by the investigator to be significantly severe; 3) grade 3 neutropenia accompanied by infection or fever of ≥38.5℃

SECONDARY OUTCOMES:
Pharmacokinetic parameters,Tmax | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  Peak time, reflecting the absorption, distribution, metabolism and excretion characteristics of drugs in the body.
Pharmacokinetic parameters, Cmax | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  Peak concentrations, reflecting the absorption, distribution, metabolism and excretion characteristics of drugs in the body.
Pharmacokinetic parameters, λz | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  The apparent terminal elimination rate constant, obtained by taking a half-log linear regression at the elimination phase concentration point, reflecting the absorption, distribution, metabolism and excretion characteristics of drugs in the body.
Pharmacokinetic parameters, t1/2 | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  the apparent terminal elimination half-life, calculated according to the following equation:t1/2= Ln(2)/ λz,reflecting the absorption, distribution, metabolism and excretion characteristics of drugs in the body.
Pharmacodynamic parameters, blood cadmium | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  blood cadmium concentration before and after drug administration
Pharmacodynamic parameters, urine cadmium | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  urine cadmium level before and after drug administration (μmol/mol creatinine)
Pharmacodynamic parameters, 24-hour urine cadmium | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  24-hour urine cadmium excretion before and after drug administration
Pharmacodynamic parameters,serum electrolyte and trace element | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  serum electrolyte and trace element concentrations before and after drug administration
Pharmacodynamic parameters, other blood heavy metals | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  whole blood heavy metal levels before and after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Fang Pei, PhD-c, Principal Investigator — Hunan Occupational Disease Prevention and Control Institute; Xiaobin Deng, Principal Investigator — Hunan Occupational Disease Prevention and Control Institute
Locations (1):
- Hunan Occupational Disease Prevention and Control Institute, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang X, Zhu J, Zhong Z, Luo M, Li G, Gong Z, Zhang C, Fei F, Ruan X, Zhou J, Liu G, Li G, Olson J, Ren X. Mobilization and removing of cadmium from kidney by GMDTC utilizing renal glucose reabsorption pathway. Toxicol Appl Pharmacol. 2016 Aug 15;305:143-152. doi: 10.1016/j.taap.2016.06.001. Epub 2016 Jun 6. PMID 27282297
- [Background] Li Guangxian. Study on the efficacy of GMDTC in removing cadmium and its toxic side effects in chronic cadmium-poisoned mice and rats [D]. Guangdong Pharmaceutical University, 2015.
- [Background] Guidelines for the management of Phase I clinical trials of drugs (trial implementation).
- [Background] Guidelines for the validation of quantitative analysis methods for biological samples in the 2020 edition of the Chinese Pharmacopoeia.